CLINICAL TRIAL: NCT05633667
Title: A Phase 2 Platform Study Evaluating the Safety and Efficacy of Novel Treatment Combinations in Patients With Lung Cancer (VELOCITY-Lung)
Brief Title: Study of Novel Treatment Combinations in Patients With Lung Cancer
Acronym: VELOCITY-Lung
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-624-6376; MOH_2022-12-13_012231 (Registry Identifier: Israel Clinical Research Site)
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer; Advanced or Metastatic Non-Small-Cell Lung Cancer; Resectable Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — zimberelimab; sacituzumab govitecan; Carboplatin; Cisplatin; Pemetrexed; Paclitaxel; 130-nm albumin-bound paclitaxel; Docetaxel; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Substudy 01: Zimberelimab (ZIM) + Sacituzumab govitecan-hziy (SG) + Domvanalimab (DOM) (Experimental): Participants will receive ZIM, SG and DOM until disease progression (PD), unacceptable toxicity, or protocol specified discontinuation criteria are met.
  Interventions: Drug: Zimberelimab (ZIM); Drug: Domvanalimab (DOM); Drug: Sacituzumab govitecan-hziy (SG)
- Substudy 01: ZIM + DOM + Etrumadenant (ETRUMA) (Experimental): Participants will receive ZIM, DOM and ETRUMA until PD, unacceptable toxicity, or protocol specified discontinuation criteria are met.
  Interventions: Drug: Zimberelimab (ZIM); Drug: Domvanalimab (DOM); Drug: Etrumadenant (ETRUMA)
- Substudy 01: ZIM + ETRUMA (Experimental): Participants will receive ZIM and ETRUMA until PD, unacceptable toxicity, or protocol specified discontinuation criteria are met.
  Interventions: Drug: Zimberelimab (ZIM); Drug: Etrumadenant (ETRUMA)
- Substudy 01: Zimberelimab (ZIM) + Sacituzumab govitecan-hziy (SG) (Experimental): Participants will receive ZIM and SG until disease progression (PD), unacceptable toxicity, or protocol specified discontinuation criteria are met.
  Interventions: Drug: Zimberelimab (ZIM); Drug: Sacituzumab govitecan-hziy (SG)
- Substudy 01: ZIM + Platinum Based Chemotherapy (Active Comparator): Expansion Stage Only: Participants will receive ZIM plus any one of the chemotherapy (choice of chemotherapy is dependent on histology).
  Platinum Based Chemotherapy will be cisplatin or carboplatin and pemetrexed (non-squamous histology) or carboplatin, paclitaxel and nabpaclitaxel (squamous histology).
  Interventions: Drug: Zimberelimab (ZIM); Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Nab-paclitaxel
- Substudy 02: SG + ZIM + ETRUMA (Experimental): Participants will receive SG, ZIM and ETRUMA until PD, unacceptable toxicity, or protocol specified discontinuation criteria are met.
  Interventions: Drug: Zimberelimab (ZIM); Drug: Sacituzumab govitecan-hziy (SG); Drug: Etrumadenant (ETRUMA)
- Substudy 02: Either Docetaxel or SG (Monotherapy Only) (Active Comparator): Participants will receive either Docetaxel or SG until PD, unacceptable toxicity, or protocol specified discontinuation criteria are met.
  Interventions: Drug: Sacituzumab govitecan-hziy (SG); Drug: Docetaxel
- Substudy 03 - ZIM + DOM + Platinum-based Chemotherapy (Experimental): Participants will receive ZIM plus DOM and any one of the chemotherapy (choice of chemotherapy is dependent on histology).
  Platinum Based Chemotherapy will be carboplatin and pemetrexed (non-squamous histology) or carboplatin and paclitaxel (squamous histology).
  Interventions: Drug: Zimberelimab (ZIM); Drug: Domvanalimab (DOM); Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel
- Substudy 03 - ZIM + Platinum-based Chemotherapy (Experimental): Participants will receive ZIM plus any one of the chemotherapy (choice of chemotherapy is dependent on histology).
  Platinum Based Chemotherapy will be carboplatin and pemetrexed (non-squamous histology) or carboplatin and paclitaxel (squamous histology).
  Interventions: Drug: Zimberelimab (ZIM); Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel
- Substudy 03: Nivolumab + Platinum-based Chemotherapy (Active Comparator): Participants will receive nivolumab plus any one of the chemotherapy (choice of chemotherapy is dependent on histology).
  Platinum Based Chemotherapy will be carboplatin and pemetrexed (non-squamous histology) or carboplatin and paclitaxel (squamous histology).
  Interventions: Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Nivolumab

INTERVENTIONS:
Drug: Zimberelimab (ZIM) — Administered intravenously
  Other Names: AB122; GS-0122
  Arms: Substudy 01: ZIM + DOM + Etrumadenant (ETRUMA); Substudy 01: ZIM + ETRUMA; Substudy 01: ZIM + Platinum Based Chemotherapy; Substudy 01: Zimberelimab (ZIM) + Sacituzumab govitecan-hziy (SG); Substudy 01: Zimberelimab (ZIM) + Sacituzumab govitecan-hziy (SG) + Domvanalimab (DOM); Substudy 02: SG + ZIM + ETRUMA; Substudy 03 - ZIM + DOM + Platinum-based Chemotherapy; Substudy 03 - ZIM + Platinum-based Chemotherapy
Drug: Domvanalimab (DOM) — Administered intravenously
  Other Names: AB154; GS-0154
  Arms: Substudy 01: ZIM + DOM + Etrumadenant (ETRUMA); Substudy 01: Zimberelimab (ZIM) + Sacituzumab govitecan-hziy (SG) + Domvanalimab (DOM); Substudy 03 - ZIM + DOM + Platinum-based Chemotherapy
Drug: Sacituzumab govitecan-hziy (SG) — Administered intravenously
  Other Names: GS-0132; IMMU-132
  Arms: Substudy 01: Zimberelimab (ZIM) + Sacituzumab govitecan-hziy (SG); Substudy 01: Zimberelimab (ZIM) + Sacituzumab govitecan-hziy (SG) + Domvanalimab (DOM); Substudy 02: Either Docetaxel or SG (Monotherapy Only); Substudy 02: SG + ZIM + ETRUMA
Drug: Etrumadenant (ETRUMA) — Administered orally
  Other Names: AB928; GS-0928
  Arms: Substudy 01: ZIM + DOM + Etrumadenant (ETRUMA); Substudy 01: ZIM + ETRUMA; Substudy 02: SG + ZIM + ETRUMA
Drug: Carboplatin — Administered intravenously
  Arms: Substudy 01: ZIM + Platinum Based Chemotherapy; Substudy 03 - ZIM + DOM + Platinum-based Chemotherapy; Substudy 03 - ZIM + Platinum-based Chemotherapy; Substudy 03: Nivolumab + Platinum-based Chemotherapy
Drug: Cisplatin — Administered intravenously
  Arms: Substudy 01: ZIM + Platinum Based Chemotherapy
Drug: Pemetrexed — Administered intravenously
  Arms: Substudy 01: ZIM + Platinum Based Chemotherapy; Substudy 03 - ZIM + DOM + Platinum-based Chemotherapy; Substudy 03 - ZIM + Platinum-based Chemotherapy; Substudy 03: Nivolumab + Platinum-based Chemotherapy
Drug: Paclitaxel — Administered intravenously
  Arms: Substudy 01: ZIM + Platinum Based Chemotherapy; Substudy 03 - ZIM + DOM + Platinum-based Chemotherapy; Substudy 03 - ZIM + Platinum-based Chemotherapy; Substudy 03: Nivolumab + Platinum-based Chemotherapy
Drug: Nab-paclitaxel — Administered intravenously
  Arms: Substudy 01: ZIM + Platinum Based Chemotherapy
Drug: Docetaxel — Administered intravenously
  Arms: Substudy 02: Either Docetaxel or SG (Monotherapy Only)
Drug: Nivolumab — Administered intravenously
  Arms: Substudy 03: Nivolumab + Platinum-based Chemotherapy

SUMMARY:
The goal of this platform clinical trial is to test how well novel treatment combinations work in participants with lung cancer. Substudy-01 will compare the different novel combinations versus standard of care in participants with metastatic (cancer that has spread) non-small-cell lung cancer (NSCLC) who have not been treated before. Substudy-02 will compare the different novel combination versus standard of care in participants with cancer that has progressed after receiving previous treatment for metastatic NSCLC. Substudy-03 will compare the different novel combinations versus standard of care in participants with resectable stage II-III NSCLC.

The primary objectives of this study are:

Substudy-01 and Substudy-02: To evaluate the objective response rate (ORR) assessed per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1).

Substudy-03: To evaluate the efficacy of treatment combinations based on complete pathological response (pCR) rate.

ELIGIBILITY:
Key Inclusion Criteria:

All Substudies:

* Histologically or cytologically documented non-small-cell lung cancer (NSCLC).
* No known actionable genomic alterations for which targeted therapies are available.
* Eastern cooperative oncology group (ECOG) performance status score of 0 or 1.
* Measurable disease per response evaluation criteria in solid tumors.
* Adequate hematologic and end-organ function.
* Individuals of childbearing potential who engage in heterosexual intercourse must agree to use specified method(s) of contraception.

Substudy 01: All Experimental arms

* Stage IV NSCLC.
* For individuals with nonsquamous histology: Epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) alteration negative.
* PD-L1 status by central confirmation.
* No prior systemic treatment for metastatic NSCLC.

Substudy 02: All Experimental arms

* Stage IV NSCLC.
* In individuals with nonsquamous histology and actionable EGFR, ALK, or other known genomic alterations must have received treatment with at least 1 targeted therapy to the appropriate genomic alteration.

Substudy 03: All Experimental arms

* Previously untreated individuals with resectable (Stage II, IIIA, IIIB (T[3-4]N2) NSCLC (per American Joint Committee on Cancer (AJCC) Edition 8).
* Planned surgery must comprise of lobectomy, sleeve lobectomy, or bi-lobectomy.
* PD-L1 status by central confirmation.
* For individuals with nonsquamous histology: Epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) alteration negative.

Key Exclusion Criteria:

All Substudies:

* Mixed small-cell lung cancer and NSCLC histology.
* Active second malignancy.
* Active autoimmune disease.
* History of or current non-infectious pneumonitis/interstitial lung disease.
* Active serious infection within 4 weeks prior to study treatment.

Substudy 01 and 02

* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Received previous anticancer therapy within 4 weeks prior to enrollment.

Substudy 03: All Experimental arms

* NSCLC previously treated with systemic therapy or radiotherapy.
* Received prior treatment with any anti-PD-(L)-1 or other immune checkpoint inhibitors (CPIs).

Note: Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 593 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Substudies 01 and 02: Objective Response Rate (ORR) as Assessed by the Investigator According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Up to 5 years
  ORR is defined as the proportion of participants achieving a complete response (CR) or partial response (PR) as confirmed at least 4 weeks after the first detection of response.
Substudy 03: Complete Pathological Response (pCR) Rate | Up to 5 years
  pCR is defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes as assessed by local pathology review.

SECONDARY OUTCOMES:
Substudies 01 and 02: Progression-free Survival (PFS) According to RECIST Version 1.1 | Up to 5 years
  PFS is defined as the time from the date of randomization until disease progression (PD) or death, whichever comes first.
Substudies 01 and 02: Duration of response (DOR) According to RECIST Version 1.1 | Up to 5 years
  DOR is defined as the time from the first response (CR or PR) until the first documented PD, or death, whichever comes first.
All Substudies: Overall survival (OS) | Up to 5 years
  OS is defined as the time from the date of randomization until death from any cause.
Substudy 03: Event-Free Survival (EFS) | Up to 5 years
  Event-Free Survival (EFS) is defined as the time from randomization until any of the following events: any progression precluding surgery or preventing completion of surgery, progression or recurrence of disease after surgery (local or distant), as assessed by investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1), or death due to any cause, whichever occurs first. Participants who do not undergo surgery for reasons other than progression will be considered to have had an event at progression or at death.
Substudy 03: Major Pathological Response (MPR) Rate | Up to 5 years
  MPR rate is defined as the percentage of participants with ≤ 10% residual tumor in lung and lymph nodes at surgery as evaluated by local pathology review.
All Substudies: Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) and Related TEAEs | First dose date up to 24 months plus 100 days
All Substudies: Percentage of Participants Experiencing Clinical Laboratory Abnormalities | First dose date up to 24 months plus 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (100):
- United States (20):
  - Arizona Oncology Associates,Substudy-01, Tucson, Arizona
  - Arizona Oncology Associates,Substudy-02, Tucson, Arizona
  - Rocky Mountain Cancer Center,Substudy-01, Denver, Colorado
  - Rocky Mountain Cancer Center,Substudy-02, Denver, Colorado
  - Fort Wayne Medical Oncology and Hematology, Inc.,Substudy-03, Fort Wayne, Indiana
  - Baptist Health Lexington,Substudy-03, Lexington, Kentucky
  - Washington University School of Medicine - Siteman Cancer Center,Substudy-01, St Louis, Missouri
  - Washington University School of Medicine - Siteman Cancer Center,Substudy-02, St Louis, Missouri
  - Washington University School of Medicine - Siteman Cancer Center,Substudy-03, St Louis, Missouri
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Oncology Hematology Care Clinical Trials, LLC,Substudy-01, Cincinnati, Ohio
  - Oncology Hematology Care Clinical Trials, LLC,Substudy-02, Cincinnati, Ohio
  - Oncology Associates of Oregon, PC,Substudy-01, Eugene, Oregon
  - Oncology Associates of Oregon, PC,Substudy-02, Eugene, Oregon
  - Texas Oncology - Central South,Substudy-01, Austin, Texas
  - Texas Oncology - Central South,Substudy-02, Austin, Texas
  - US Oncology Investigational Products Center (IPC),Substudy-01, Fairfax, Virginia
  - US Oncology Investigational Products Center (IPC),Substudy-02, Fairfax, Virginia
  - Fred Hutchinson Cancer Center,Substudy-01, Seattle, Washington
  - Fred Hutchinson Cancer Center,Substudy-02, Seattle, Washington
- Brazil (10):
  - Fundação Pio XII - Hospital de Amor,Substudy-01, Barretos
  - Centro Gaúcho Integrado de Oncologia Hematologia, Ensino e Pesquisa Ltda./Hospital Mãe de Deus,Substudy-03, Porto Alegre
  - Hospital Mae de Deus,Substudy-01, Porto Alegre
  - Hospital Mae de Deus, Porto Alegre
  - Hospital Sao Lucas da PUC Rio Grande do Sul,Substudy-01, Porto Alegre
  - Hospital Sao Lucas da PUC Rio Grande do Sul,Substudy-03, Porto Alegre
  - BP-A Beneficencia Portuguesa De Sao Paulo,Substudy-01, São Paulo
  - Fundação Antonio Prudente - Hospital do Câncer AC Camargo,Substudy-01, São Paulo
  - Fundação Antonio Prudente/A.C. Camargo Cancer Center,Substudy-03, São Paulo
  - Real e Benemérita Associação Portuguesa de Beneficência/Hospital Beneficência Portuguesa de São Paulo (Hospital BP),Substudy-03, São Paulo
- Hong Kong (6):
  - Queen Mary Hospital,Substudy-01, Hong Kong
  - Queen Mary Hospital,Substudy-02, Hong Kong
  - Queen Elizabeth Hospital,Substudy-01, Hong Kong
  - Queen Elizabeth Hospital,Substudy-02, Hong Kong
  - Prince of Wales Hospital,Substudy-01, New Territories
  - Prince of Wales Hospital,Substudy-02, New Territories
- Israel (12):
  - Rambam Health Care Campus,Substudy-01, Haifa
  - Rambam Health Care Campus,Substudy-02, Haifa
  - Rambam Health Care Campus,Substudy-03, Haifa
  - Shaare Zedek Medical Center,Substudy-01, Jerusalem
  - Shaare Zedek Medical Center,Substudy-02, Jerusalem
  - Shaare Zedek Medical Center,Substudy-03, Jerusalem
  - Hadassah Medical Center,Substudy-01, Jerusalem
  - Hadassah University Medical Center,Substudy-03, Jerusalem
  - Rabin Medical Center,Substudy-03, Petah Tikva
  - Tel Aviv Sourasky Medical Center,Substudy-01, Tel Aviv
  - Tel Aviv Sourasky Medical Center,Substudy-02, Tel Aviv
  - Tel-Aviv Sourasky Medical Center,Substudy-03, Tel Aviv
- South Korea (24):
  - Chungbuk National University Hospital,Substudy-01, Cheongju-si
  - Chungbuk National University Hospital,Substudy-02, Cheongju-si
  - National Cancer Center,Substudy-01, Goyang
  - National Cancer Center,Substudy-02, Goyang
  - National Cancer Center,Substudy-03, Goyang
  - Chonnam National University Hwasun Hospital,Substudy-01, Gwangju
  - Chonnam National University Hwasun Hospital,Substudy-03, Gwangju
  - Seoul National University Bundang Hospital,Substudy-01, Gyeonggi-do
  - Seoul National University Bundang Hospital,Substudy-03, Gyeonggi-do
  - Kosin University Gospel Hospital,Substudy-01, Seogu
  - Kosin University Gospel Hospital,Substudy-03, Seogu
  - Severance Hospital, Yonsei University Health System,Substudy-03, Seoul
  - Asan Medical Center,Substudy-02, Seoul
  - Asan Medical Center,Substudy-03, Seoul
  - Asan Medical Centre,Substudy-01, Seoul
  - Samsung Medical Center,Substudy-01, Seoul
  - Samsung Medical Center,Substudy-02, Seoul
  - Samsung Medical Center,Substudy-03, Seoul
  - Severance Hospital, Yonsei University Health System,Substudy-01, Seoul
  - Severance Hospital, Yonsei University Health System,Substudy-02, Seoul
  - Seoul National University,Substudy-01, Seoul
  - Seoul National University,Substudy-02, Seoul
  - Korea University Guro Hospital,Substudy-01, Seoul
  - Korea University Guro Hospital,Substudy-03, Seoul
- Taiwan (11):
  - Changhua Christian Hospital,Substudy-01, Changhua
  - Changhua Christian Hospital,Substudy-02, Changhua
  - Changhua Christian Hospital,Substudy-03, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital,Substudy-01, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital,Substudy-02, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital,Substudy-03, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital,Substudy-01, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital,Substudy-02, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital,Substudy-03, Kaohsiung City
  - National Taiwan University Hospital,Substudy-01, Taipei
  - National Taiwan University Hospital,Substudy-02, Taipei
- Turkey (Türkiye) (10):
  - Adana City Training and Research Hospital,Substudy-01, Adana
  - Memorial Ankara Hastanesi,Substudy-01, Ankara
  - Memorial Ankara Hospital,Substudy-03, Ankara
  - Medical Park Samsun,Substudy-01, Atakum
  - Dicle University,Substudy-01, Diyarbakır
  - Dicle University Medical Faculty,Substudy-03, Diyarbakır
  - Necmettin Erbakan University Meram Faculty of Medicine,Substudy-01, Konya
  - Necmettin Erbakan Universitesi,Substudy-03, Meram Konya
  - Gazi University Medical Faculty,Substudy-01, Yenimahalle
  - Gazi University Medical Faculty,Substudy-03, Yenimahalle
- United Kingdom (7):
  - Birmingham Heartlands Hospital,Substudy-03, Birmingham
  - University Hospitals Birmingham NHS Trust,Substudy-01, Birmingham
  - University Hospitals Birmingham NHS Trust,Substudy-02, Birmingham
  - St James University Hospital,,Substudy-01, Leeds
  - St. Bartholomew's Hospital,Substudy-01, London
  - St. Bartholomew's Hospital,Substudy-02, London
  - St. Bartholomew's Hospital,Substudy-03, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-624-6376